CLINICAL TRIAL: NCT02277808
Title: Which Apparatus for Inhaled Pentamidine? A Comparison of Drug Delivery to the Lung Between Two Nebulizers: The Respirgard II and the Isoneb.
Brief Title: Which Apparatus for Inhaled Pentamidine?
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, G.Reychler, Doctor in Physiotherapy, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Nebulizers for pentamidine
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: Pneumocystis; Nebulizer; Pentamidine
MeSH Terms: conditions — Pneumonia, Pneumocystis | interventions — Amikacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Respirgard II (Active Comparator): Determination of pulmonary deposition
  Interventions: Drug: 500mg Amikacine (Amukin®) diluted in 4mL NaCl (0,9%); Device: Respirgard II
- Isoneb (Active Comparator): Determination of pulmonary deposition
  Interventions: Drug: 500mg Amikacine (Amukin®) diluted in 4mL NaCl (0,9%); Device: Isoneb®

INTERVENTIONS:
Drug: 500mg Amikacine (Amukin®) diluted in 4mL NaCl (0,9%)
Device: Respirgard II
  Arms: Respirgard II
Device: Isoneb®
  Arms: Isoneb

SUMMARY:
The reference nebulizer used for pentamidine nebulization is currently the Respirgard II ®, disposable pneumatic nebulizer. Other nebulizers are on the market and appear to have comparable properties and better availability to the hospital. Several studies remark that all nebulizers with comparable properties could be used for the nebulization.The aim of our work will be to evaluate and compare the pulmonary deposition between the reference nebulizer Respirgard II ®, and one of these nebulizers available on the market, the Isoneb ®. We will measure and compare these data's for each of the nebulizers via nebulization Amikacine and urinary dosage.

ELIGIBILITY:
Inclusion Criteria:

* Be in good health

Exclusion Criteria:

* Known Tachycardia
* Renal Dysfunction
* Respiratory Diseases and history

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Amikacine urinary dosage | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Grégory Reychler, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Clinique universitaire Saint-Luc, Brussels, Belgium

REFERENCES:
- [Background] Oudyi M, Chaumuzeau JP, Diot P, Dubus JC; GAT (Groupe Aerosoltherapie de la SPLF). [Use of pentamidine nebulization in children]. Rev Mal Respir. 2012 May;29(5):656-63. doi: 10.1016/j.rmr.2012.02.003. Epub 2012 Mar 28. French. PMID 22682591
- [Background] McIvor RA, Berger P, Pack LL, Rachlis A, Chan CK. An effectiveness community-based clinical trial of Respirgard II and Fisoneb nebulizers for Pneumocystis carinii prophylaxis with aerosol pentamidine in HIV-infected individuals. Toronto Aerosol Pentamidine Study (TAPS) Group. Chest. 1996 Jul;110(1):141-6. doi: 10.1378/chest.110.1.141. PMID 8681618
- [Background] Kim CS, Garcia L, Wanner A. Actual pentamidine dose delivered by Respigard II nebulizer. Eur Respir J. 1995 Dec;8(12):2178-81. doi: 10.1183/09031936.95.08122178. PMID 8666114